CLINICAL TRIAL: NCT01186523
Title: Long-term Exercise, Weight Loss and Energy Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Joseph Donnelly, Professor, University of Kansas
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSCL15226; R01DK049181 (NIH)
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
Keywords: Obesity; Weight Management; Physical Activity
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 400 kcal of exercise/session (Experimental): 400 kcal of exercise/session
  Interventions: Other: Long Term Energy Balance
- 600 Kcal of exercise/session (Experimental): 600 Kcal of exercise/session
  Interventions: Other: Long Term Energy Balance
- Control, no exercise (Experimental): No exercise control group
  Interventions: Other: Long Term Energy Balance

INTERVENTIONS:
Other: Long Term Energy Balance — To see if there is a variance in weight loss and energy balance between men and women with similar energy expenditure over an extended period of time.
  Other Names: 400 kcal of exercise/session; 600 kcal of exercise/session; No exercise control group

SUMMARY:
In order to examine potential gender differences in the weight loss response to exercise, the investigators propose to compare equal energy expenditure of exercise for overweight men and women using levels of exercise energy expenditure that the investigators have previously shown to prevent weight gain or promote weight loss. The investigators will randomize men and women to an exercise group, 5 days/week, for 9 months, with an energy expenditure of 400 kcal/exercise session, a group with 600 kcal/ exercise session, or a control group. 1)The investigators hypothesize that men and women randomized to sedentary control will gain weight, those randomized to 400 kcal/exercise session will maintain weight (will not gain), and those randomized to 600 kcal/exercise session will lose ~5% of body weight. 2) The investigators hypothesize there will be no differences for weight loss between genders at either 400 or 600 kcal of energy expenditure of exercise since men and women will have equal amounts of energy expenditure of exercise. 3) The investigators hypothesize that men and women randomized to 400 kcal/exercise session will completely compensate for the energy expended during exercise by altering energy intake and/or spontaneous activity and that men and women participants randomized to 600 kcal/exercise session will not completely compensate. The investigators believe the findings from this study could have important implications for exercise guidelines for weight loss.

DETAILED DESCRIPTION:
Exercise is recommended by virtually every public health organization; however, the role of exercise is generally considered secondary to energy restriction for the treatment of obesity. Indeed, an argument can be made that suggests exercise is not effective for weight loss. Meta-analytic studies consistently find small amounts of weight loss due to exercise without energy restriction. It is critical to note that there are actually very few randomized controlled trials using exercise alone for weight loss. We believe that there are 3 critical flaws in the vast majority of the literature. 1)Participants are not supervised and is generally recorded by self report and is likely poorly estimated and in general, overestimated. 2)The amount of exercise used is usually prescribed from the guidelines for recommended levels for physical fitness and to diminish cardiovascular disease, not the amount that may be necessary for weight loss. 3)The energy expenditure of the exercise is rarely reported.

Participants will be randomly assigned to expend either 400 or 600kcal per exercise session (or a control group) and will exercise 5 days per week for 9 months. All exercise sessions will be supervised and the length of the exercise session will be based upon energy expenditure (kcal/min) at a give heart rate range. To account for improvements in fitness, energy expenditure will be measured monthly and adjustments to the daily exercise prescription will be altered accordingly.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or greater
* males & females
* <500kcal exercise/wk
* BMI 25-40

Exclusion Criteria:

* known cardiovascular and metabolic disorders,
* weight altering product use
* smoking
* clinical depression
* special diets

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2005-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Between group weight change at 10 months | 10 months

SECONDARY OUTCOMES:
Body Composition | 10 months
  Changes in body composition will be evaluated by measuring the change in percent body fat, total fat mass, and total lean mass by DEXA.
Resting Metabolic Rate | 10 months
  Resting metabolic rate will be determined via indirect calorimetry following an overnight fast.
Total Daily Energy Expenditure | 10 months
  Total daily energy expenditure will be determined using the doubly labeled water procedure

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Donnelly, EdD, Principal Investigator — University of Kansas
Locations (1):
- Energy Balance Lab, The University of Kansas, Lawrence, Kansas, United States

REFERENCES:
- [Derived] Herrmann SD, Willis EA, Honas JJ, Lee J, Washburn RA, Donnelly JE. Energy intake, nonexercise physical activity, and weight loss in responders and nonresponders: The Midwest Exercise Trial 2. Obesity (Silver Spring). 2015 Aug;23(8):1539-49. doi: 10.1002/oby.21073. PMID 26193059
- [Derived] Ptomey LT, Willis EA, Honas JJ, Mayo MS, Washburn RA, Herrmann SD, Sullivan DK, Donnelly JE. Validity of energy intake estimated by digital photography plus recall in overweight and obese young adults. J Acad Nutr Diet. 2015 Sep;115(9):1392-9. doi: 10.1016/j.jand.2015.05.006. Epub 2015 Jun 26. PMID 26122282
- [Derived] Donnelly JE, Honas JJ, Smith BK, Mayo MS, Gibson CA, Sullivan DK, Lee J, Herrmann SD, Lambourne K, Washburn RA. Aerobic exercise alone results in clinically significant weight loss for men and women: midwest exercise trial 2. Obesity (Silver Spring). 2013 Mar;21(3):E219-28. doi: 10.1002/oby.20145. PMID 23592678